CLINICAL TRIAL: NCT03616041
Title: Video Capsule Endoscopy for Lesion Localization and Diagnosis in Patients With Severe Hematochezia
Brief Title: Capsule Endoscopy for Severe Hematochezia
Status: Recruiting | Type: Observational
Sponsor: CURE Digestive Diseases Research Center (Other)
Responsible Party: Principal Investigator, Dennis M Jensen, M.D., Professor of Medicine, CURE Digestive Diseases Research Center
Other Study IDs: Colon Capsule
Record Dates: First submitted 2018-07-16; First posted 2018-08-06 (Actual); Last update posted 2024-08-12 (Actual); Status verified 2024-08

CONDITIONS: Hematochezia
Keywords: Severe hematochezia
MeSH Terms: conditions — Gastrointestinal Hemorrhage

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

GROUPS / COHORTS (1):
- Colon capsule endoscopy: Participant who meet the eligible criteria undergo an evaluation for severe hematochezia with a second-generation colon capsule endoscopy system in addition to standard diagnostic tests including tagged RBC scan, and/or computerized tomographic angiography (CTA), and/or conventional angiography.
  Interventions: Device: Second-generation colon capsule endoscopy system

INTERVENTIONS:
Device: Second-generation colon capsule endoscopy system — The PillCam (TM) Colon 2 which is a second-generation colon capsule endoscopy system, developed by Medtronic Inc. Colon capsule endoscopy, in contrast to current generation small bowel capsules, is capable of visualizing the entire lumen and mucosa from esophagus to rectum. This can be crucial for patients being screened or evaluated for colon disorders. This new generation of colon capsule endoscopy has a battery life of at least 10 hours and preserves energy using adaptive frame rate technology.

SUMMARY:
Patients with severe hematochezia (bright red blood per rectum) may have a bleeding source proximal to the colon. Visualization of the entire gastrointestinal tract using a second-generation colon capsule endoscopy system could improve diagnostic yields and form the basis for a new approach to early diagnosis that could change guidelines and practice management in these patients. The hypothesis of this study is that urgent colon capsule endoscopy will have higher rates of lesion localization and diagnosis and reduced time to diagnosis than the standard tagged red blood cell scanning and/or angiography. In this study, the eligible patients with severe hematochezia are enrolled to undergo an evaluation with the capsule endoscopy in addition to the standard tests including a tagged RBC scan and/or an angiogram. The outcomes in terms of diagnostic yields of the capsule endoscopy will be compared to the standard tests.

DETAILED DESCRIPTION:
Background and Significance

Currently there are no consensus guidelines for the best approach to patient with severe hematochezia. One strategy is to perform an urgent colonoscopy (following a colon purge) within 12-15 hours. Although this strategy has been associated with a decreased length of hospitalization and an improved diagnostic and therapeutic yields, it has drawbacks. A major disadvantage of performing an urgent colonoscopy is that the endoscopist can evaluate only the colon and the distal ileum, while more proximal sources of bleeding are not evaluated. Another limitation is that thorough cleansing of the colon is required to facilitate complete evaluation, identification of stigmata of recent hemorrhage and lesion diagnosis. Urgent colonoscopy is labor intense and relies on a dedicated bleeding team with expertise in both diagnosis and hemostasis. Another option for patients with persistent or recurrent hematochezia is to perform either a tagged RBC scan or an angiogram to identify the bleeding location. However, these techniques also have major disadvantages, including low diagnostic yields for severe hematochezia, requiring additional tests for diagnosis, and cannot visually detect non-bleeding stigmata of hemorrhage on lesions that can be seen during colonoscopy or by capsule endoscopy.

Research Design and Methods This is a study of patients who being admitted to the hospital for severe hematochezia or inpatients who developed hematochezia after hospitalization for an unrelated non-GI bleeding reason. Those who meet entry criteria and lack exclusions on screening before will being asked to participate in this study.

After informed consent, patients will be a colon preparation prior to ingestion of the colon capsule. The capsule recording system will be activated once patients swallow the capsule. Once the capsule has been excreted or if the capsule stops recording images (usually 10 hours after activation), the video recorder will then be taken to a workstation and the video will be downloaded for reading.

In addition to having the capsule endoscopy, all consented patients will undergo standard tests for the initial diagnosis and management of severe hematochezia: tagged RBC scan and/or computerized tomographic angiography (CTA), magnetic resonance imaging (MRI) angiogram, or conventional angiography. Because of contra indication, MRI angiography will not be performed until the capsule has been excreted, nor will CT angiography because the capsule may interfere with interpretation. All patients will also have urgent colonoscopy after clearing the colon of blood and stool with the purge. All of these diagnostic procedures will be performed within 48 hours of GI consultation, but ideally as soon as possible.

If a bleeding site is not identified by colonoscopy, further diagnostic workup are usually performed as part of the standard of care, including anoscopy, esophagogastroduodenoscopy, push enteroscopy, or deep enteroscopy. If bleeding continues or worsens, surgery may be necessary to control the bleeding.

The GI endoscopist, nuclear medicine physician, and radiologist will be blinded to the results of the capsule endoscopy until 24 hours after the other diagnostic tests (i.e. tagged RBC scan, angiography, and endoscopy/colonoscopy) have been performed. Then the results of all tests will be unblinded. This will be done for the purpose of not delaying clinical management, but also to avoid biasing the interpretations of these diagnostic studies.

Data Collection and Monitoring Demographic data and medical history including details of co-morbid illnesses, risk factors, and characteristics of the GI bleeding will be recorded. Reasons for exclusion will be documented. Baseline physical examinations, American Society of Anesthesiology (ASA) classification, laboratory results, Blatchford-Glasgow score, units of blood products transfused, and results of the real-time viewer will also be recorded. Results of RBC scanning, angiography, capsule endoscopy, endoscopy, pathology, and surgery will be recorded. The outcomes including rates of re-bleeding or persistent bleeding, treatment of bleeding at endoscopy or radiology, need for surgery, major complications, transfusions after initial resuscitation, hospital and intensive care unit days, and death will be prospectively recorded up to the time of hospital discharge and 30 days following discharge. Subgroup analysis regarding results of urgent colonoscopy/enteroscopy will be performed to assess for differences in diagnostic yield and therapeutic interventions between different endoscopists. The number of patients who experience any difficulties in capsule swallowing will be recorded, including inability to swallow the capsule, incomplete examination of small bowel or colon, and capsule retention.

Sample size calculation The initial sample size estimate was made from results of our prior comparative retrospective study of small bowel capsule endoscopy in patients with severe hematochezia. In that study, the diagnostic yield of tagged red blood cell scanning and/or CTA was 47% and the urgent capsule endoscopy was 67%. For 80% power to detect a 20% difference in diagnostic yield at a 0.05 level, a sample size of 46 patients was calculated. Accounting for patients who consented but had incomplete testing, 14 additional patients would be enrolled for a total of 60 patients.

Based upon actual May 2022 preliminary results of 11 patients who were hospitalized with severe hematochezia and completed the diagnostic testing with both standard imaging and colon capsule, a revised study sample size was estimated. This was based upon a diagnostic yield of RBC scanning or angiography of 25 % and the diagnostic yield of colon capsule of 75% for patients with severe hematochezia. With this 50% difference in diagnostic yield (for both bleeding site localization and lesion diagnosis), 19 total patients would yield statistically significant results. This is with a very conservative estimate for an alpha of 0.05 and 90% power - a beta of 0.10 with two-tailed testing. Including those patients who consented but have incomplete testing, we propose a total enrollment of 23 patients. This is a new sample size to complete the study.

Statistical analysis methods A descriptive analysis will be performed for baseline demographic characteristics. Continuous data will be summarized as means ± standard deviations and categorical data will be summarized as percentages. The primary end point of the study will be the diagnostic yield (defined as the frequency of detection and percentage of positive results) for each technique for the localization of the bleeding site and/or etiologic diagnosis (e.g. definitive if stigmata of recent hemorrhage are found or presumptive if a clean lesion is diagnosed and no other lesions are found by complete evaluation). The diagnostic yield of each technique will be calculated and compared by the McNemar test for paired data using exact methods. The sensitivity, specificity, and accuracy will be determined for lesion localization; absence of lesions in the foregut, small bowel, or colon; and etiologic diagnosis (definitive or presumptive) for capsule endoscopy, tagged red blood cell scan/angiography, and endoscopy. The final diagnosis by endoscopy, angiography, pathology, and surgery will be considered the gold standard. Concordance between each diagnostic strategy will be calculated and reported with the kappa index. A p-value of less than 0.05 will be considered statistically significant.

Confidentiality:

Study data will be physically and electronically secured. All personal information will be replaced with a code de-identifying subject's information. The researchers will do their best to make sure that all subject's private information is kept confidential as possible.

Data Management Records will be labelled with a code number and then only de-identified information will be entered into our encrypted Statistical Analysis System (SAS) electronic database located at the VA West Los Angeles. No identifiable information about them will be kept in the electronic research data files. All personal information will be replaced with a code. A list linking the code and their identifiable information will be kept separate from the research data files in a locked file in the research team's office located at VA West Los Angeles. (VA CURE GI Hemostasis Research Unit). This list will be protected by the Principal Investigator (Dennis Jensen, MD) and the research team. At the end of the study, the investigators will destroy this link and no one - not even the researchers - will be able to connect their identity to the research data.

Future Use of Data After the study finishes, the research team will continue to use the patient's de-identified medical data from their medical history, laboratory results, labs, radiological, surgical, and pathology results, and colonoscopy results and information on their medical progress to continue to analyze and to report new GI research results.

Data and Safety Monitoring Plan

Adverse events The following adverse event information will be prospectively collected: capsule retention rates and those requiring endoscopic removal, perforations, aspiration, myocardial infarctions, strokes, and deaths within 30 days of enrollment.

Frequency Safety data will be collected daily while hospitalized and weekly after discharge from the hospital, up to 30 days after enrollment. Data collection will start as soon as the patient enrolls in the study and swallows the capsule.

Review Cumulative safety data will be reviewed every 30 days.

All serious adverse events (SAE's) will be reported to the IRB as mandated by the VA research service.

The safety data will be overseen by the PI and the biostatistician. All results will be reported to the IRB, who will review all SAE's.

Based upon widespread utilization and safety of capsule endoscopy for small bowel bleeding since 2001 in the U.S. and many other countries worldwide, the investigators do not expect any clinical condition which would trigger an immediate suspension of this research study.

ELIGIBILITY:
Inclusion Criteria:

1. 18 years old or older
2. Able to provide written informed consent or have a legal surrogate who can provide written consent
3. Presenting with evidence of severe ongoing hematochezia (i.e. passage of red blood or clots per rectum witnessed by a health care provider) and have a decrease in hemoglobin from baseline of 2 or more grams and/or transfusion of 1 or more units of red blood cells for resuscitation with either outpatient or inpatient start of severe hematochezia.

Exclusion Criteria:

1. Uncooperative, unable to give written informed consent personally or through a legal surrogate, or refuse to participate
2. Contraindication to undergo capsule endoscopy due to:

   1. Documented or suspected bowel obstruction (partial or complete)
   2. Anatomical GI abnormalities such as strictures of the foregut or small bowel
   3. Inability to swallow the capsule
   4. Presence of cardiac pacemakers or other implanted electromedical devices
3. American Society of Anesthesiology (ASA) class V (very severe co-morbidities and very poor prognosis for surgery or similar procedures)
4. Very severe GI bleeding with shock not responsive to IV fluid resuscitation and/or transfusions and IV medications to raise the systolic blood pressure
5. History of recent hematemesis (within 30 days), positive nasogastric, or orogastric (OG) aspirate suggesting an upper GI bleed
6. Presenting with recurrent hematochezia that has been previously diagnosed as anorectal bleeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients who are hospitalized with severe GI bleeding (hematochezia) thought to be from a colonic or small bowel source, who meet entry criteria and lack exclusions.
Sampling Method: Non-Probability Sample
Enrollment: 23 (Estimated)
Dates: Start 2021-02-10 (Actual); Primary Completion 2024-10-30 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
The diagnostic yield tests in detecting a bleeding site and comparison of rates | 30 days
  The diagnostic yield of the bleeding site detection (defined as the rates of detection and percentage of positive results as eg. positive test or total tests) for capsule endoscopy, tagged red blood cell scan/angiography, and endoscopy will be calculated. Rates of positive detection will be compared by the McNemar test for data using exact methods.

SECONDARY OUTCOMES:
The sensitivity for lesion localization | 30 days
  The sensitivity for lesion localization for capsule endoscopy, tagged red blood cell scan/angiography, and endoscopy will be calculated and compared.
The specificity for lesion localization | 30 days
  The specificity for lesion localization for capsule endoscopy, tagged red blood cell scan/angiography, and endoscopy will be calculated and compared.
The accuracy for lesion localization | 30 days
  The accuracy for lesion localization for capsule endoscopy, tagged red blood cell scan/angiography, and endoscopy will be calculated and compared.

CONTACTS AND LOCATIONS:
Overall Officials: Dennis M. Jensen, MD, Principal Investigator — VA Greater Los Angeles Healthcare System
Locations (2):
- United States (2):
  - VA Greater Los Angeles Healthcare System, Los Angeles, California
  - Ronald Reagan UCLA Medical Center, Los Angeles, California

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Strate LL. Lower GI bleeding: epidemiology and diagnosis. Gastroenterol Clin North Am. 2005 Dec;34(4):643-64. doi: 10.1016/j.gtc.2005.08.007. PMID 16303575
- [Background] Lanas A, Garcia-Rodriguez LA, Polo-Tomas M, Ponce M, Alonso-Abreu I, Perez-Aisa MA, Perez-Gisbert J, Bujanda L, Castro M, Munoz M, Rodrigo L, Calvet X, Del-Pino D, Garcia S. Time trends and impact of upper and lower gastrointestinal bleeding and perforation in clinical practice. Am J Gastroenterol. 2009 Jul;104(7):1633-41. doi: 10.1038/ajg.2009.164. Epub 2009 May 5. PMID 19574968
- [Background] Camus M, Khungar V, Jensen DM, Ohning GV, Kovacs TO, Jutabha R, Ghassemi KA, Machicado GA, Dulai GS. Origin, Clinical Characteristics and 30-Day Outcomes of Severe Hematochezia in Cirrhotics and Non-cirrhotics. Dig Dis Sci. 2016 Sep;61(9):2732-40. doi: 10.1007/s10620-016-4198-y. Epub 2016 Jun 10. PMID 27286877
- [Background] Zuckerman GR, Prakash C. Acute lower intestinal bleeding. Part II: etiology, therapy, and outcomes. Gastrointest Endosc. 1999 Feb;49(2):228-38. doi: 10.1016/s0016-5107(99)70491-8. No abstract available. PMID 9925703
- [Background] Jensen DM, Machicado GA. Colonoscopy for diagnosis and treatment of severe lower gastrointestinal bleeding. Routine outcomes and cost analysis. Gastrointest Endosc Clin N Am. 1997 Jul;7(3):477-98. PMID 9177148
- [Background] Jensen DM, Machicado GA, Jutabha R, Kovacs TO. Urgent colonoscopy for the diagnosis and treatment of severe diverticular hemorrhage. N Engl J Med. 2000 Jan 13;342(2):78-82. doi: 10.1056/NEJM200001133420202. PMID 10631275
- [Background] Jensen DM, Ohning GV, Kovacs TO, Jutabha R, Ghassemi K, Dulai GS, Machicado GA. Natural history of definitive diverticular hemorrhage based on stigmata of recent hemorrhage and colonoscopic Doppler blood flow monitoring for risk stratification and definitive hemostasis. Gastrointest Endosc. 2016 Feb;83(2):416-23. doi: 10.1016/j.gie.2015.07.033. Epub 2015 Jul 31. PMID 26227931
- [Background] Kanwal F, Dulai G, Jensen DM, Gralnek IM, Kovacs TO, Machicado GA, Jutabha R. Major stigmata of recent hemorrhage on rectal ulcers in patients with severe hematochezia: Endoscopic diagnosis, treatment, and outcomes. Gastrointest Endosc. 2003 Apr;57(4):462-8. doi: 10.1067/mge.2003.147. PMID 12665754
- [Background] Jensen DM. Management of patients with severe hematochezia--with all current evidence available. Am J Gastroenterol. 2005 Nov;100(11):2403-6. doi: 10.1111/j.1572-0241.2005.00298.x. PMID 16279892
- [Background] Spada C, Hassan C, Munoz-Navas M, Neuhaus H, Deviere J, Fockens P, Coron E, Gay G, Toth E, Riccioni ME, Carretero C, Charton JP, Van Gossum A, Wientjes CA, Sacher-Huvelin S, Delvaux M, Nemeth A, Petruzziello L, de Frias CP, Mayershofer R, Amininejad L, Dekker E, Galmiche JP, Frederic M, Johansson GW, Cesaro P, Costamagna G. Second-generation colon capsule endoscopy compared with colonoscopy. Gastrointest Endosc. 2011 Sep;74(3):581-589.e1. doi: 10.1016/j.gie.2011.03.1125. Epub 2011 May 20. PMID 21601200
- [Background] Boal Carvalho P, Rosa B, Dias de Castro F, Moreira MJ, Cotter J. PillCam COLON 2 in Crohn's disease: A new concept of pan-enteric mucosal healing assessment. World J Gastroenterol. 2015 Jun 21;21(23):7233-41. doi: 10.3748/wjg.v21.i23.7233. PMID 26109810
- [Background] Camus M, Jensen DM, Ohning GV, et al. Urgent capsule endoscopy for bleeding site localization & lesion diagnosis of patients with severe hematochezia. Gastrointest Endosc 2013;77: AB274